CLINICAL TRIAL: NCT03521960
Title: Buspirone as an Adjunctive Medication for Opioid Tapering
Brief Title: Buspirone for Opioid Tapering
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00125620
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Opioid-Related Disorders; Dependency (Psychology); Pain, Chronic; Opiate Withdrawal Syndrome
Keywords: Buspirone
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Buspirone

STUDY DESIGN:
Intervention Model Description: Patient completing a residential stay on the Pain Treatment Unit in which this study is being conducted will be enrolled and randomly assigned to receive either buspirone or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind placebo controlled study. Patients are randomized to receive either active buspirone or placebo, each of which is over-encapsulated to support blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buspirone oral capsule (Active Comparator): Buspirone (15 milligrams) administered orally three times per day
  Interventions: Drug: Buspirone oral capsule
- Placebo oral capsule (Placebo Comparator): Placebo administered orally three times per day
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Buspirone oral capsule — 15 milligrams, three times daily
  Other Names: Buspar
  Arms: Buspirone oral capsule
Drug: Placebo oral capsule — 0 milligrams (placebo), three times daily
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
This is a pilot study to collect preliminary data to support a grant application. The goal of the study is to evaluate whether the Food and Drug Administration (FDA)-approved and generically-available medication buspirone reduces symptoms of opioid withdrawal among patients undergoing a clinically-indicated and supervised taper from their opioid pain medications. This is premised on strong preclinical scientific support but has not yet be well-examined in humans.

DETAILED DESCRIPTION:
Buspirone (Buspar) has shown initial efficacy in reducing symptoms of opioid withdrawal in animal studies and in human patients undergoing a methadone taper. Buspirone may have pharmacologic activity in specific neurotransmitter systems that preclinical evidence suggests may be implicated in the manifestation of opioid withdrawal symptoms. Administration of buspirone during an opioid taper may improve outcomes relative to placebo. The goal of this study is to collect preliminary feasibility and efficacy data from a sample of patients undergoing clinically-indicated opioid tapering. Participant enrollment will occur at the beginning of their residential stay on the Pain Treatment Unit at Johns Hopkins Hospital. Participants will be randomly assigned to receive buspirone (15 milligrams, three times daily, for daily dose of 45 milligrams) or placebo. Daily assessments for withdrawal and requests for additional symptomatic medications will be evaluated as evidence of initial efficacy. Feasibility measures include willingness to participate and study retention.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Be undergoing taper of prescribed opioid pain medications at the study site

Exclusion Criteria:

* Being pregnant or breastfeeding
* Past 7-day use of grapefruit juice or other strong Cytochrome (CYP) P450 inhibitors or inducers
* Have medical or psychiatric condition that is contraindicated with buspirone administration
* Current suicidality as assessed by clinic staff or the Columbia Suicide Severity Rating Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Taper Completion | 28 days
  Final day on which participant is enrolled in the clinic
Opioid Withdrawal Symptom Severity | 28 days
  Daily ratings of the Subjective Opiate Withdrawal Scale (SOWS)Total Score. The SOWS is a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely), and takes less than 10 minutes to complete.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT03521960/Prot_SAP_000.pdf